CLINICAL TRIAL: NCT00960271
Title: Medico-economic Evaluation of a Preoperative Algorithm Including EBUS for NSCLC Initial Staging
Brief Title: Evaluation of Preoperative Endobronchial Ultrasound (EBUS) in Non Small Cell Lung Cancer (NSCLC)
Acronym: EVIEPEB
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2007/138/HP; EVIEPEB
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non-small cell lung cancer; mediastinal lymph node; resectable; EBUS; stage IIIA; significant mediastinal lymph node at thoracic CT Scan
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- NON SMALL CELL LUNG CANCER: Non small cell lung cancer, with clinical N2 disease, otherwise operable.
  Interventions: Procedure: EBUS

INTERVENTIONS:
Procedure: EBUS — a minimally invasive technique of mediastinal lymph node staging using an integrated videoendoscopic device equipped with ultrasound for the localization and transbronchial sampling of lymph nodes in real time
  Other Names: NSCLC

SUMMARY:
This study aims to assess both the role and cost-effectiveness of EBUS in preoperative Non small cell lung cancer staging. This controlled multicentric study will be conducted in 22 centers in France. The study design includes two prospective phases. In phase 1, one investigator in each center will prospectively be evaluated for its ability to perform EBUS, with a required goal of 9 informative samplings out of 10 consecutive patients. The phase 2 will include the medico-economic assessment of the technique in the preoperative setting. A maximum of 420 patients for each phase is forecasted.

ELIGIBILITY:
Inclusion Criteria:

* adult patients over 18
* non small cell lung cancer histologically or cytologically proved
* Clinical Stage IIIA
* anatomically and functionally resectable

Exclusion Criteria:

* uncorrected bleeding disorders
* absence of lymphadenopathy superior to 1cm in small axis at CT scan
* contraindication to bronchoscopy
* extrathoracic or intrathoracic metastasis
* respiratory function tests not compatible with curative resection of lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include non small cell lung cancer patients, stage III A (before PET Scan), with resectable tumors.
Sampling Method: Non-Probability Sample
Enrollment: 363 (Actual)
Dates: Start 2008-09; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
number of mediastinoscopy avoided | 24h

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital, Rouen, France

REFERENCES:
- [Derived] Chouaid C, Salaun M, Gounant V, Febvre M, Vergnon JM, Jouniaux V, Fournier C, Lachkar S, Hermant C, Raspaud C, Quantin X, Quiot JJ, Molard A, Dayen C, Marquette CH, Lena H, Zalcman G, Thiberville L. Clinical efficacy and cost-effectiveness of endobronchial ultrasound-guided transbronchial needle aspiration for preoperative staging of non-small-cell lung cancer: Results of a French prospective multicenter trial (EVIEPEB). PLoS One. 2019 Jan 7;14(1):e0208992. doi: 10.1371/journal.pone.0208992. eCollection 2019. PMID 30615623